CLINICAL TRIAL: NCT05948891
Title: Impact of Fixed TRIple Therapy With Beclometasone/Formoterol/Glycopyrronium DPI (Trimbow® in NEXThaler Device) in Chronic Obstructive PulmoNary Disease in rEal-world Settings: Health-related Quality of Life Patient' eXpectations and characterisTics: the TriNEXT Study
Acronym: TriNEXT
Status: Recruiting | Type: Observational
Sponsor: Chiesi SAS (Industry)
Collaborators: Kappa Santé (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS 723
Record Dates: First submitted 2023-06-30; First posted 2023-07-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: COPD
Keywords: Digital; QOL; PROMS; PRO; respiratory diseases; Chronic obstructive pulmonary disease (COPD); Adult; observational; connected device; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases | interventions — Beclomethasone; Formoterol Fumarate; Glycopyrrolate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Beclometasone/Formoterol/Glycopyrronium 88 µg/5 µg/9 µg DPI (Trimbow® 88 µg/5 µg/9 µg in NEXThaler device) — observational, prospective, multicentric, international, cohort study

SUMMARY:
This is an observational, prospective, multicentric, cohort study conducted in France to evaluate the QoL in COPD patients treated with TRIMBOW NEXThaler 88/5/9 in a routine clinical practice setting. Patients enrolled in this study will be patients diagnosed with a COPD with a ratio of post-bronchodilator (salbutamol 400 μg) forced expiratory volume in 1 s (FEV1) to forced vital capacity (FVC) of less than 0.7 to whom TRIMBOW NEXThaler 88/5/9 has been initiated by an hospital or local pulmonologists in accordance with clinical practice and marketing authorization.

DETAILED DESCRIPTION:
The decision of patients to participate in this study must not, in any way, impact upon the standard of care that they are receiving or any benefits to which they are otherwise entitled. The treatment decision must have been taken prior to and independently of the patient's inclusion in the study. All aspects of treatment and clinical management of patients will be at the discretion of the participating pulmonologist (or treating pulmonologist where different) according to local clinical practice and applicable local regulations.

In addition to the data available per clinical practice, the participating pulmonologists will be asked to obtain patient-reported outcome measures (PROMs) data from patients within this study and to invite patients to wear a connected watch to record physical activity and sleep quality (50% of patients (about 250 patients) who first accept to wear the watch will be equipped).

The duration of a patient's participation in this study will be 6 months made of three visits (M0, M3, M6) according to routine clinical practice.

* Visit 1 (M0); inclusion of patient when BDP/FF/GB NEXThaler® 88/5/9 is initiated;
* Visit 2 (M3); 3 months (+/- 30 days) post BDP/FF/GB NEXThaler® 88/5/9 initiation;
* Visit 3 (M6, last visit): 6 months (+/- 30 days) post BDP/FF/GB NEXThaler® 88/5/9 initiation;

The inclusion duration will be 12 to 15 months. The overall duration of the study, including recruitment and follow-up, is expected to be 21 months.

Data collection will be considered complete for a participating patient if data available at 6 have been recorded in the CRF and associated PROs completed. Patients will be followed until the end of the study period (M6) even if TRIMBOW NEXThaler 88/5/9 is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥40 years
* Diagnosis of COPD with a ratio of post-bronchodilator (salbutamol 400 μg) forced expiratory volume in 1 s (FEV1) to forced vital capacity (FVC) of less than 0.7
* Physicians' decision to start a first prescription fixed triple therapy with BDP/FF/GB NEXThaler® 88/5/9 in accordance with the marketing authorization
* COPD Assessment Test (CAT) total score of at least 10 at the day of inclusion
* Informed consent to participate in the study

Exclusion Criteria:

* Asthmatic patients
* Patients with moderate or severe exacerbations within the 4 weeks prior to enrolment
* Patients treated with fixed triple therapies within 6 months prior inclusion
* Patients receiving pulmonary rehabilitation within 3 months prior to inclusion or within 6 months after inclusion
* Concomitant participation in experimental clinical studies/investigations or participation in experimental clinical studies/investigations within 3 months prior to enrolment into the present study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participating in this non-interventional real-world evidence study will be COPD patients for whom it has been decided to initiate BDP/FF/G (88/5/9) in NEXThaler® device by a physician in accordance with clinical practice
  All eligible patients should be offered enrolment for data collection within the study. Participating sites will be encouraged to propose the study to all patients satisfying eligibility criteria, in a consecutive manner, when patients come for their regular consultation, in order to minimize bias in patient selection. In any case, the treatment decision must have been taken by the investigator prior to, and independently of the patient's inclusion into the study, following standard clinical practice and regulations.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change of quality of life through CAT (COPD assessement tool) over 6 month period | Month 6
  To assess change in QoL using the CAT scale over a 6-month follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device
  • Primary endpoint is the proportion of patients achieving a ≥2-point reduction in CAT total score (MCID) at M6 compared to baseline.

SECONDARY OUTCOMES:
Mean change Quality of life through VQ11 questionnaire | Month 0, Month 3 and Month 6
  To assess change in QoL using the VQ11 scale over a 6-month follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device
  • Endpoint is mean VQ11 total score and sub scores described at baseline, M3 and M6
Proportion of patients achieving a ≥2-point reduction in VQ11 total score | Month 0, Month 3 and Month 6
  To assess change in QoL using the VQ11 scale over a 6-month follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device
  • Endpoint is the proportion of patients achieving a ≥2-point reduction in VQ11 total score (MCID) at M3 and M6 compared to baseline.
Mean change in Dyspnoea throught "Dyspnea-12 questionnaire" | Month 0, Month 3 and Month 6
  To assess changes in dyspnoea using the Dyspnea-12 over a 6-month follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device
  • Endpoint is D-12 total score and sub scores described at baseline, M3 and M6
Proportion of patients achieving a 3-point reduction in "Dyspnea-12" total score | Month 0, Month 3 and Month 6
  To assess changes in dyspnoea using the Dyspnea-12 over a 6-month follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device
  • Endpoint is the proportion of patients achieving a 3-point reduction in D-12 total score (MCID) at M3 and M6 compared to baseline.
Rate of moderate and severe exacerbations at M0, M3 and M6 through eCRF | Month 0, Month 3 and Month 6
  To describe the occurrence of moderate to severe exacerbations over a 6- month follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device
  Endpoint is the proportion of patients with at least a moderate or severe exacerbation (overall and in each category), at baseline (in the previous 12 months), M3 and M6
Proportion of patients achieving an increase in physical activity throught the a connected device | Month 0, Month 3 and Month 6
  To assess changes in physical activity using a connected watch over a 6-month
  • Endpoint is the proportion of patients achieving an increase in physical activity (≥ 10%-increase in the mean daily number of step) at M3 and M6 compared to baseline.
  Baseline physical activity (M0) will be defined as the mean of data collected during the first 7 days of connected device wearing watch over a 6-month follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device
Mean daily number of steps throught the a connected device | Month 0, Month 3 and Month 6
  To assess changes in physical activity using a connected watch over a 6-month
  • Endpoints are the mean daily number of steps and the mean of number of steps during 7 days at M0, M3 and M6
  Baseline physical activity (M0) will be defined as the mean of data collected during the first 7 days of connected device wearing watch over a 6-month follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device
Sleep quality throught the Pittsburgh questionnaire | Month 0, Month 3 and Month 6
  • Endpoints are the Pittsburgh questionnaire at M0, M3 and M6
  Baseline physical activity (M0) will be defined as the mean of data collected during the first 7 days of connected device wearing.
Sleep quality throught the a connected device | Month 0, Month 3 and Month 6
  To assess changes in sleep quality using a connected device
  • Endpoints are the mean daily sleep time, the mean of sleep time and the mean daily number of awakenings during 7 days at M0, M3 and M6
  Baseline sleep quality (M0) will be defined as the mean of data collected during the first 7 days of connected device wearing.
Treatment compliance at M3 and M6 through TAI (test inhaler adherence) questionnary | Month 3 and Month 6
  To assess treatment compliance with BDP/FF/G (88/5/9) in NEXThaler® device
  • Endpoint is the description of treatment compliance global score at M3 and M6 for COPD using TAI
Baseline description of sociodemographic data and medical data through eCRF | baseline
  to describe COPD patient, disease and treatment characteristics at initiation of BDP/FF/G (88/5/9) in NEXThaler® device
  * Endpoints are description of sociodemographic (age, sex, weight, height, education level, occupation), medical data (risk factors exposure including tobacco, disease history) and lung function data (FEV1, FVC, RV, TLC) at baseline
  * Endpoints are description of comorbidities and associated treatment throughout the study at baseline
  * Endpoints are description of previous COPD-related treatment at baseline through eCRF
Treatment tolerance throughout the study through eCRF | up to 24 weeks
  To assess treatment tolerance in COPD patients treated with with BDP/FF/G (88/5/9) in NEXThaler® device To assess patient satisfaction with treatment in COPD patients treated with BDP/FF/GB NEXThaler® 88/5/9

OTHER OUTCOMES:
Correlation between exacerbations occurrence and physical activity | Month 6
  To assess the association between exacerbations occurrence and physical activity changes
  Physical activity measured by a connected device over a 6-month follow-up
Correlation between exacerbations occurrence and sleep quality | Month 6
  To assess the association between exacerbations occurrence sleep quality changes
  Sleep quality changes measured by a connected device over a 6-month follow-up period in COPD patients treated with BDP/FF/G (88/5/9) in NEXThaler® device for COPD
Correlation between QoL measured by VQ11 and the CAT through PROM | Month 0, Month 3 and Month 6
  To assess the correlation between QoL measured with the VQ11 and the CAT for COPD
  • Endpoints are value of the Pearson correlation test described at baseline, M3 and M6
Correlation between QoL measured with the VQ11 and Dyspnea-12 through PROM | Month 0, Month 3 and Month 6
  To assess the correlation between QoL measured with the VQ11 and Dyspnea-12 for COPD
  • Endpoints are value of the Pearson correlation test described at baseline, M3 and M6
Among patients with the connected device, assess the correlation of sleep quality when measured with connected device and with the Pittsburgh Sleep Quality Index | Month 0, Month 3 and Month 6
  Among COPD patients with the connected device, to assess the correlation of sleep quality when measured with connected device and with the Pittsburgh Sleep Quality Index
  • Endpoints are value of the Pearson correlation test described at baseline, M3 and M6
Dyspnoea with modified Medical Research Council (mMRC) | Month 0, Month 3 and Month 6
  Endpoint is mMRC total score described at baseline, M3 and M6

CONTACTS AND LOCATIONS:
Overall Officials: Capucine MORELOT PANZINI, Pr, Principal Investigator — University Hospital, la pitié salpêtrière; Philippe DEVILLIER, Pr, Principal Investigator — HOSPITAL, FOCH; Hervé PEGLIASCO, Dr, Principal Investigator — European Hospital, Marseille
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided